CLINICAL TRIAL: NCT04819009
Title: Can the Enhanced Transtheoretical Model Intervention (ETMI) be Implemented in a Public Health Organization- an Implementation Study
Brief Title: Can the Enhanced Transtheoretical Model Intervention (ETMI) be Implemented in a Public Health Organization
Status: Completed | Type: Observational
Sponsor: Ariel University (Other)
Collaborators: Maccabi Healthcare Services, Israel (Other)
Responsible Party: Sponsor
Other Study IDs: ArielURF
Record Dates: First submitted 2021-03-18; First posted 2021-03-26 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2023-01

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; implementation study; Enhanced Transtheoretical Model Intervention; Public Health
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Central District: The ETMI method will be implemented in this group
  Interventions: Other: the Enhanced Transtheoretical Model Intervention (ETMI)
- North District: control
- Hasharon District: control
- South District: control
- Jerusalem and Hasfhela District: control

INTERVENTIONS:
Other: the Enhanced Transtheoretical Model Intervention (ETMI) — ETMI consists of a physical and functional examination, a discussion about the role of physical activity matched to the patient stage of change, and guided through motivational interviewing techniques, exposure to fast walking, and goal setting. The patient receives a postcard outlining the main messages about physical activity and four simple stretches.
  The ETMI method consists of four parts:
  1. Creating a therapeutic alliance (communication skills and reassurance)
  2. Clear messages to the patient: Mandatory 3 sentences: (1." physical activity is the only thing that will help your back pain over time." 2. "It's easy to reduce your pain now - but the important thing is to prevent the next episode"," 3. "Your body must be strong and flexible.")
  3. Exposure to brisk walking (brisk walking in the corridor, hand by hand with the therapist) and graded activity.
  4. Postcard with reminder messages on how to self manage the back.
  Groups: Central District

SUMMARY:
The aim of this study is to assess whether the ETMI method can be implemented among primary care practitioners in the central district of Maccabi Health Services and examine whether it provides a medical and economic advantage.

DETAILED DESCRIPTION:
An implementation study- a prospective cohort study with pre- and post-intervention by retrieving economic and therapeutic outcome data from MHS databases. The intervention group will be the Central District of MHS, among 220 primary care practitioners (100 Physicians and 120 physiotherapists) and their patients (n=7,000) who suffer from back pain and receive treatment. We will investigate the relationship between the care received and outcomes in terms of healthcare utilization, costs, and patient-relevant outcomes.

ELIGIBILITY:
Inclusion Criteria:

* primary care practitioners and their patients, who suffer from back pain and receive treatment.
* patients who suffer from back pain and receive treatment with or without leg radiation

Exclusion Criteria:

* no

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 220 primary care practitioners (100 Physicians and 120 physiotherapists) and their patients (n=7,000) who suffer from back pain and receive treatment.
Sampling Method: Non-Probability Sample
Enrollment: 1463 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
ETMI Code | baseline

SECONDARY OUTCOMES:
Lumbar Computerized Adaptive Test (LCAT) | baseline
  LCAT is a computerized adaptive test, meaning that the administration selects items from the item bank one at a time based on an administrative algorithm. The final calculated functional score ranges on a linear scale of 0-100, higher measures representing higher function. Additionally, the system predicts a risk-adjusted functional score at discharge. The adjusting is on: functional score at admission, age, sex, chronicity as number of days from onset of the treated condition, number of related surgeries, exercise history and use of medication to treat LBP.MCID for the LCAT is 3-9 points depending on the first score. LCAT has been tested for validity by comparing it to the Oswestry Low Back Pain Disability Questionnaire and has a high level of reliability in the English version (α = 0.92).Several studies have been published using the LCAT's Hebrew version.

OTHER OUTCOMES:
Economic variables and therapeutic results | baseline
  Number of primary care clinician appointments
Numeric Pain Rate Scale (NPRS) | baseline
  The patient is asked to rate his pain intensity in the last 24 hours on a scale of 0-10 (10=severest pain)
Fear Avoidance Belief Questionnaire (FABQ) | baseline
  It is a modification to the original version, allowing for the assessment using an Item Response Theory-based measures replacing the summative methods. The later version consists of three items, scoring 0-100, with 100 representing higher fear-avoidance, and 44 being a cut-off point between high and low values
Economic variables and therapeutic results | baseline
  Number of orthopedic clinician appointments
Economic variables and therapeutic results | baseline
  Number of physiotherapy appointments
Economic variables and therapeutic results | baseline
  Anti-inflammatory drug dosage
Economic variables and therapeutic results | baseline
  Number of imaging tests
Economic variables and therapeutic results | baseline
  Number of surgeries and procedures

CONTACTS AND LOCATIONS:
Overall Officials: Ron Feldman, PhD Candidate, Principal Investigator — Ariel University
Locations (1):
- Ariel University, Ariel, Israel

IPD SHARING:
Plan to Share IPD: Yes
the result of the study will be analyzed. a paper will be submitted to an international journal with study description including methods, examination protocol results.
Supporting Information: Study Protocol, CSR
Time Frame: one year following completion of study

REFERENCES:
- [Background] Ben-Ami N, Chodick G, Mirovsky Y, Pincus T, Shapiro Y. Increasing Recreational Physical Activity in Patients With Chronic Low Back Pain: A Pragmatic Controlled Clinical Trial. J Orthop Sports Phys Ther. 2017 Feb;47(2):57-66. doi: 10.2519/jospt.2017.7057. PMID 28142364
- [Background] Canaway A, Pincus T, Underwood M, Shapiro Y, Chodick G, Ben-Ami N. Is an enhanced behaviour change intervention cost-effective compared with physiotherapy for patients with chronic low back pain? Results from a multicentre trial in Israel. BMJ Open. 2018 Apr 10;8(4):e019928. doi: 10.1136/bmjopen-2017-019928. PMID 29643158
- [Background] Simoneau GG. 2017 JOSPT Award Recipients. J Orthop Sports Phys Ther. 2018 May;48(5):348. doi: 10.2519/jospt.2018.0104. PMID 29712542